CLINICAL TRIAL: NCT02427165
Title: A Phase II, Randomised, Double Blind, Placebo Controlled, Seven Way Crossover Study to Assess the Effect of Single Doses of RPL554 Compared to Salbutamol and Placebo Administered by Nebuliser on Lung Function of Patients With Chronic Asthma
Brief Title: Comparison of RPL554 With Placebo and Salbutamol in Asthmatic Patients
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Verona Pharma plc (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Treatment
Other Study IDs: RPL554-008-2014
Record Dates: First submitted 2015-04-14; First posted 2015-04-27 (Estimated); Last update posted 2016-09-09 (Estimated); Status verified 2016-09

CONDITIONS: Asthma
MeSH Terms: conditions — Asthma | interventions — ensifentrine; Albuterol

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (7):
- Placebo (Placebo Comparator): Single dose of nebulised placebo solution
  Interventions: Drug: Placebo
- RPL554 Dose 1 (Experimental): 0.4 mg single dose nebulised RPL554
  Interventions: Drug: RPL554
- RPL554 Dose 2 (Experimental): 1.5 mg single dose nebulised RPL554
  Interventions: Drug: RPL554
- RPL554 Dose 3 (Experimental): 6 mg single dose nebulised RPL554
  Interventions: Drug: RPL554
- RPL554 Dose 4 (Experimental): 24 mg single dose nebulised RPL554
  Interventions: Drug: RPL554
- Salbutamol Dose 1 (Active Comparator): 2.5 mg single dose nebulised salbutamol
  Interventions: Drug: Salbutamol
- Salbutamol Dose 2 (Active Comparator): 7.5 mg single dose nebulised salbutamol
  Interventions: Drug: Salbutamol

INTERVENTIONS:
Drug: RPL554 — A dual PDE3 and PDE4 inhibitor
  Other Names: VMX554; VRP554
  Arms: RPL554 Dose 1; RPL554 Dose 2; RPL554 Dose 3; RPL554 Dose 4
Drug: Salbutamol — a beta-2 receptor agonist
  Arms: Salbutamol Dose 1; Salbutamol Dose 2
Drug: Placebo — RPL554 placebo containing no active ingredients
  Arms: Placebo

SUMMARY:
The number of people with of asthma and allergy is still increasing and a large number of patients still do not have their asthma well controlled. There is therefore a need for new asthma treatments that work well and have less side effects. The study compares a new experimental drug RPL554 with a marketed asthma drug (salbutamol) and placebo.

DETAILED DESCRIPTION:
A seven way crossover study to investigate the pharmacodynamics, pharmacokinetics, safety and tolerability of inhaled RPL554 compared to salbutamol and placebo in patients with mild to moderate chronic asthma.

Salbutamol is a marketed beta-2 agonist typically used to treat bronchospasm (due to any cause, allergen asthma or exercise-induced), as well as chronic obstructive pulmonary disease but has associated dose-related systemic side effects.

RPL554 is a dual PDE3 and PDE4 inhibitor that has bronchodilatory and anti-inflammatory actions and also the potential to stimulate increases in mucociliary clearance via its proven ability to activate CFTR. Four different doses of RPL554 will be compared with placebo and a two doses of salbutamol as benchmarks for bronchodilation and systemic side effects.

ELIGIBILITY:
Inclusion Criteria:

* Provided written informed consent
* Males agree not to donate sperm and either be abstinent or use adequate contraception. Females to be post-menopausal or surgically sterile
* Non-smoker or ex-smoker >6 months
* Diagnosed asthma for at least 6 months
* Pre-bronchodilator FEV1 ≥60% and ≤90% of predicted normal value and ≥1.5 L at screening
* Increase in FEV1 of 15% within 30 minutes after a 2.5mg dose of nebulised salbutamol
* Systolic blood pressure 90 to 145 mmHg, diastolic blood pressure 50 to 90 mmHg and heart rate 45 to 80 beats per minute (bpm) after resting for 5 minutes in a supine position (average from two measurements)
* Capable of withdrawing from LABAs, LAMAs and SAMAs before screening and during study and SABAs before screening and for 8 hours before each dose

Exclusion Criteria:

* Asthma exacerbation in the last 3 months
* Any prior life threatening episode of asthma (intensive care admission)
* Any clinically significant disease or disorder or clinically relevant screening result
* QTcF interval >450 ms or QT interval >500 ms or other abnormality in ECG
* History of ischemic heart disease or heart failure. History of recurrent or current clinically significant arrhythmia or ECG abnormality as judged by the investigator
* Treatment with systemic glucocorticosteroids within 30 days before screening
* A suspected/manifested infection according to WHO risk classification 2, 3 or 4

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 29 (Actual)
Dates: Start 2015-04; Primary Completion 2015-11 (Actual); Study Completion 2015-11 (Actual)

PRIMARY OUTCOMES:
Spirometry | 12 hours
  FEV1

SECONDARY OUTCOMES:
Spirometry | 4, 6 and 8 hours
  FEV1
Systemic pharmacodynamic effect on blood pressure | 4 hours
  Supine blood pressure in the 4 hours after nebulisation
Systemic pharmacodynamic effect on pulse rate | 4 hours
  Supine Pulse rate in the 4 hours after nebulisation
Systemic pharmacodynamic effect on ECG heart rate | 4 hours
  ECG heart rate in the 4 hours after nebulisation
Vital signs (Supine pulse rate) | 12 hours
  Supine pulse rate
Vital signs (Supine blood pressure) | 12 hours
  Supine systolic and diastolic blood pressure
ECG | 12 hours
  12-lead ECG parameters
Pharmacokinetics (AUC) | 12 hours
  RPL554 AUC
Pharmacokinetics (Cmax) | 12 hours
  RPL554 Cmax
Pharmacokinetics (tmax) | 12 hours
  RPL554 tmax
Pharmacokinetics (half life) | 12 hours
  RPL554 half life
Pharmacokinetics (MRT) | 12 hours
  RPL554 MRT

CONTACTS AND LOCATIONS:
Overall Officials: Lief Bjermer, Principal Investigator — Skane University Hospital, Sweden; Johnston Stewart, Principal Investigator — Celerion, Northern Ireland
Locations (2):
- Skane University Hospital, Lund, Sweden
- Celerion, Belfast, United Kingdom

REFERENCES:
- [Derived] Bjermer L, Abbott-Banner K, Newman K. Efficacy and safety of a first-in-class inhaled PDE3/4 inhibitor (ensifentrine) vs salbutamol in asthma. Pulm Pharmacol Ther. 2019 Oct;58:101814. doi: 10.1016/j.pupt.2019.101814. Epub 2019 Jun 14. PMID 31202957